CLINICAL TRIAL: NCT05450978
Title: Physiological-based Pharmacokinetics Approach to Determine the Extent of Drug Exposure of Antiseizure Medications During Pregnancy and Breastfeeding
Brief Title: Physiological-based Pharmacokinetics Approach to Medication Exposure During Pregnancy and Breastfeeding
Acronym: PBPK
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Page B. Pennell, MD, Professor, University of Pittsburgh
Other Study IDs: STUDY21090138; R01HD105305 (NIH)
Record Dates: First submitted 2022-06-22; First posted 2022-07-11 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy; Pregnancy Related
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine; Levetiracetam; Oxcarbazepine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood, urine, breast milk, umbilical cord blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lamotrigine (LTG): Participants will include women with epilepsy planning pregnancy or in the early first trimester of pregnancy and treated with lamotrigine (LTG)
  Interventions: Drug: Lamotrigine
- Levetiracetam (LEV): Participants will include women with epilepsy planning pregnancy or in the early first trimester of pregnancy and treated with Levetiracetam (LEV)
  Interventions: Drug: Levetiracetam
- Oxcarbazepine (OXC): Participants will include women with epilepsy planning pregnancy or in the early first trimester of pregnancy and treated with with Oxcarbazepine (OXC)
  Interventions: Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Lamotrigine — Anti-seizure concentrations
  Other Names: Anti-seizure medication: Lamotrigine (LTG)
  Groups: Lamotrigine (LTG)
Drug: Levetiracetam — Anti-seizure concentrations
  Other Names: Anti-seizure medication: Levetiracetam (LEV)
  Groups: Levetiracetam (LEV)
Drug: Oxcarbazepine — Anti-seizure concentrations
  Other Names: Anti-seizure medication: Oxcarbazepine (OXC)
  Groups: Oxcarbazepine (OXC)

SUMMARY:
This project focuses on anti-seizure medication (ASM) clearance and physiological factors determining blood concentrations in pregnant adult women with epilepsy and amounts of exposure to their unborn children and nursing infants.

DETAILED DESCRIPTION:
The goal of this study is to develop modeling of pharmacokinetic changes for Antiseizure medications (ASMs), lamotrigine (LTG), and levetiracetam (LEV) during pregnancy and postpartum that can be used to:

1. Adjust doses in practice without obtaining frequent visits to the lab for therapeutic drug monitoring.
2. Predict exposure of ASMs in mothers and their infants in order to maintain the individualized target concentrations, thus protecting mothers from seizure worsening and minimizing fetal toxicity.

Hypotheses:

1. Drug concentrations obtained in preconception and early pregnancy predict clearance changes throughout the remainder of pregnancy for individual pregnant women with epilepsy.
2. Validated model allows the prediction of drug concentration changes at all stages throughout and after pregnancy, which will more accurately predict increased seizures and medication side effects.

Additionally, pilot data will be obtained for oxcarbazepine (OXC) in a small number of participants and contribute to data for ASMs that undergo glucuronidation (LTG).

ELIGIBILITY:
Inclusion Criteria:

* Woman with epilepsy between the ages of 18-45 planning pregnancy or in the early first trimester of pregnancy.
* Women with epilepsy ability to maintain a daily medical diary
* Women with epilepsy ability to answer side effect questionnaires
* Women with epilepsy currently being treated with lamotrigine (LTG) or levetiracetam (LEV) or oxcarbazepine (OXC)

Exclusion Criteria:

* Women with epilepsy having history of functional seizures.
* Women with epilepsy history of other major medical illnesses including renal or hepatic disease, progressive cerebral disease,
* Women with epilepsy who have inability to maintain a seizure and medication daily diary
* Women with epilepsy with present or recent history of drug or alcohol abuse, or the use of any concomitant medications that interact with the ASM they are taking (lamotrigine, levetiracetam, oxcarbazepine).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with Epilepsy
Study Population: Participants to be mainly recruited from Neurology and OBGYN clinics.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Anti-Seizure Medication (ASM) Clearance | Through study completion, an average of 18 months.
  ASM Clearance will be calculated from measurements of lamotrigine, oxcarbazepine, and levetiracetam blood concentrations, serum creatinine and 24-hour urine collection (for levetiracetam), glucuronidated metabolite (for lamotrigine), steroid hormones, medication formulation and doses, time since recent doses, and participant weight.

SECONDARY OUTCOMES:
Seizure Frequency | Through study completion, an average of 18 months.
  Participants will keep a daily seizure diary throughout their participation in the study. The diary will be reviewed at each study visit.
Anti-seizure Medication (ASM) Side Effects | Through study completion, an average of 18 months
  An ASM Side Effect Questionnaire will be administered and a neurologic examination will be performed at each study visit.
Placental passage of Anti-Seizure Medications (ASM) | Through study completion, an average of 18 months
  Maternal blood will be drawn and umbilical cord blood will be collected, for measurements of ASM concentrations for lamotrigine, oxcarbazepine, and levetiracetam.

CONTACTS AND LOCATIONS:
Overall Officials: Page B Pennell, MD, Principal Investigator — The University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will adhere to the NIH Grants Policy Statement on Sharing of Biomedical Research Resources, including the "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources: Final Notice." The results of the studies proposed here will be shared with the scientific community on a regular basis through presentations at scientific meetings and peer-reviewed publications in appropriate scientific journals. Any material resources developed as a result of this grant will be made available to other investigators once a Material Transfer Agreement has been signed between the University of Pittsburgh, University of Minnesota and the requesting investigator's institution.

REFERENCES:
- [Background] Pennell PB, French JA, May RC, Gerard E, Kalayjian L, Penovich P, Gedzelman E, Cavitt J, Hwang S, Pack AM, Sam M, Miller JW, Wilson SH, Brown C, Birnbaum AK, Meador KJ; MONEAD Study Group. Changes in Seizure Frequency and Antiepileptic Therapy during Pregnancy. N Engl J Med. 2020 Dec 24;383(26):2547-2556. doi: 10.1056/NEJMoa2008663. PMID 33369356
- [Background] Birnbaum AK, Meador KJ, Karanam A, Brown C, May RC, Gerard EE, Gedzelman ER, Penovich PE, Kalayjian LA, Cavitt J, Pack AM, Miller JW, Stowe ZN, Pennell PB; MONEAD Investigator Group. Antiepileptic Drug Exposure in Infants of Breastfeeding Mothers With Epilepsy. JAMA Neurol. 2020 Apr 1;77(4):441-450. doi: 10.1001/jamaneurol.2019.4443. PMID 31886825
- [Background] Pennell PB, Karanam A, Meador KJ, Gerard E, Kalayjian L, Penovich P, Matthews A, McElrath TM, Birnbaum AK; MONEAD Study Group. Antiseizure Medication Concentrations During Pregnancy: Results From the Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) Study. JAMA Neurol. 2022 Apr 1;79(4):370-379. doi: 10.1001/jamaneurol.2021.5487. PMID 35157004

DOCUMENTS (2):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT05450978/Prot_000.pdf
  • Informed Consent Form (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT05450978/ICF_001.pdf